CLINICAL TRIAL: NCT05147883
Title: The Effect of Exercise on Quality of Life, Sleep Quality and Anxiety in Patients With Prediabetes (EFEXQULS)
Acronym: EFEXQULS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Principal Investigator, Elif Yıldırım Ayaz, Principal Investigator, Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EFEXQULS
Record Dates: First submitted 2021-11-23; First posted 2021-12-07 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: PreDiabetes; Physical Inactivity; Quality of Life; Sleep; Anxiety; Depression
Keywords: PreDiabetes; Physical Inactivity; Quality of Life; Sleep; Anxiety; Depression
MeSH Terms: conditions — Prediabetic State; Sedentary Behavior; Anxiety Disorders; Depression | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): Patients will be given an aerobic exercise program for 1 hour, 3 days a week for 12 weeks.
  Interventions: Behavioral: Exercise
- Control (No Intervention): No intervention will be applied to the patients

INTERVENTIONS:
Behavioral: Exercise — Patients will be given an aerobic exercise program for 1 hour, 3 days a week for 12 weeks
  Arms: Exercise

SUMMARY:
The aim of this study is to determine the effect of exercise on quality of life, sleep quality and anxiety in patients with prediabetes.

DETAILED DESCRIPTION:
Randomized controlled studies are needed to examine the effects of exercise on sleep quality, quality of life, anxiety and depression in patients with prediabetes.

The aim of this study is to determine the effect of exercise on quality of life, sleep quality and anxiety in patients with prediabetes.

ELIGIBILITY:
Inclusion Criteria:

* 18-59 years old
* Living a sedentary life (physical activity below 300 kcal/day will be evaluated with the Minnesota Leisure Physical Activity Questionnaire)
* Those who have sufficient motivation to participate in the exercise program (will be evaluated by a one-on-one interview by the researchers)
* Those diagnosed with prediabetes by oral glucose tolerance test and/or HbA1c measurement will be included.
* Being eligible to participate in an exercise program after a cardiac examination (resting ECG and questioning of cardiac symptoms, advanced tests such as exercise ECG test if necessary) performed by the physician

Exclusion Criteria:

* Serious medical condition (for example, advanced malignancy or major neurological, psychiatric or endocrine disease, respiratory failure, etc.) that would prevent the person from participating in exercise training.
* Having cardiovascular disease
* Being diabetic
* Receiving hormone replacement therapy
* Life expectancy less than 1 year
* HIV positivity
* Substance use
* Functional dependency
* Cognitive weakness
* Those who have other diseases that will affect the results of the study (respiratory diseases, muscle diseases, etc.)
* Those who use drugs or supplements that will affect the results of the study

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — 18-59 years
Enrollment: 90 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Score of Quality of Life | 1 week
  Quality of Life evaluated with Health-Related Short Form-36 Survey(Min-Max:0-100). High score idicates high quality of life.

SECONDARY OUTCOMES:
Sleep Quality | 1 week
  Sleep Quality evaluated with Pitssburgh Sleep Quality Index (PSQI) (Min-max: 0-100). High score indicates worse sleep quality.
Anxiety | 1 week
  Anxiety evaluated with Hospital Anxiety Depression Scale (HADS) (Min-max:0-21). high score indicates high anxiety.
Depression | 1 week
  Depression evaluated with Hospital Anxiety Depression Scale (HADS). (Min-max:0-21). high score indicates high depression.

CONTACTS AND LOCATIONS:
Overall Officials: Elif Yıldırım Ayaz, M.D., Principal Investigator — Sultan Abdülhamid Training And Research Hospital
Locations (1):
- Sultan Abdülhamid Training and Research Hospital, Istanbul, Uskudar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No